CLINICAL TRIAL: NCT03070223
Title: Pitavastatin to REduce Physical Function Impairment and FRailty in HIV (PREPARE)
Brief Title: PREPARE (A5361s) Ancillary Study of REPRIEVE (A5332)
Acronym: PREPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTG A5361s; UM1AI068636 (NIH); R01AG054366 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — pitavastatin

STUDY DESIGN:
Intervention Model Description: Participants were randomized as part of REPRIEVE.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pitavastatin (Experimental): Participants who were randomized to pitavastatin in the main study REPRIEVE.
  Interventions: Drug: Pitavastatin
- Placebo (Placebo Comparator): Participants who were randomized to placebo for pitavastatin in the main study REPRIEVE.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pitavastatin — One tablet (4 mg) taken once daily, orally with or without food for the entire time participant was in REPRIEVE follow-up.
  Arms: Pitavastatin
Drug: Placebos — One tablet taken once daily, orally with or without food for the entire time participant was in REPRIEVE follow-up.
  Arms: Placebo

SUMMARY:
Aging with HIV is associated with earlier development of frailty (weakness) or disability, including loss of physical and muscle strength, and walking speed. Few treatments have been shown to prevent or slow these impairments in people with or without HIV. Some studies have suggested that the class of drugs called statins (for example, pitavastatin) might be helpful in slowing frailty or disability. This might happen by decreasing fat within the muscle or by decreasing inflammation markers (substances in the blood that determine how the body reacts to infection or irritation) in the blood. Other studies have shown that statins increase the risk of muscle aches and pains. This ancillary study was done to determine the impact of the drug pitavastatin on physical and muscle function.

DETAILED DESCRIPTION:
The Randomized Trial to Prevent Vascular Events in HIV (REPRIEVE (A5332), subsequently referred to as REPRIEVE; NCT02344290) was a prospective, randomized, placebo-controlled, multicenter phase III trial to evaluate pitavastatin as prevention for cardiovascular disease events among people with HIV. PREPARE (A5361s, subsequently referred to as PREPARE) was an ancillary study of REPRIEVE to determine the effects of pitavastatin on physical and muscle function. The study enrolled participants:

1. enrolled in both REPRIEVE and its Mechanistic Substudy (A5333s, subsequently referred to as Mechanistic Substudy) within 24 of their REPRIEVE enrollment
2. enrolled in REPRIEVE alone concurrently with their REPRIEVE enrollment.

The target sample size was 600 participants. The study was conducted at the REPRIEVE U.S. sites participating in the Mechanistic Substudy, and enrollment from the Mechanistic Substudy was prioritized to maximize the number of participants with computed tomography (CT) scan data performed as part of the Mechanistic Substudy.

Treatment groups (pitavastatin vs placebo) were defined according to randomization in REPRIEVE. Participants were enrolled into PREPARE blinded to their REPRIEVE treatment allocation. No intervention was provided in this ancillary study.

Originally the study duration was 48 months after participants' REPRIEVE entry. An additional visit was added at Month 60 due to missed in-person evaluations during the COVID-19 related restrictions in 2020 through early 2021.

Study visits were scheduled at PREPARE entry and at months 12, 24, 36, 48 and 60 after REPRIEVE entry. Each study visit included evaluation of physical function, frailty and self-reported physical activity and sedentary time. In addition, demographic and clinical data, laboratory specimens and CT scans collected as part of the main study REPRIEVE or its Mechanistic Substudy were used.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory participants enrolled in both REPRIEVE (A5332) and its Mechanistic Substudy (A5333s) or ambulatory participants who are newly enrolling into REPRIEVE (A5332) at A5333s ACTG sites.

Exclusion Criteria:

* Inability to ambulate independently (use of a cane or a walker is permitted) or rise from a chair without assistance.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Brown, MD, PhD, Study Chair — Johns Hopkins University; Kristine Erlandson, MD, Study Chair — University of Colorado, Denver
Locations (31):
- United States (30):
  - Alabama CRS (31788), Birmingham, Alabama
  - University of Southern California (1201), Los Angeles, California
  - University of California, Los Angeles CARE Center CRS (601), Los Angeles, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - 2701 Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Johns Hopkins University CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital (MGH) CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (31786), Newark, New Jersey
  - Weill Cornell Chelsea CRS (7804), New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU -Chelsea (7803), New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hospital (TMH) ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Trinity Health and Wellness Center CRS (31443), Dallas, Texas
  - Houston AIDS Research Team (HART) CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, PR, Puerto Rico

REFERENCES:
- [Result] Erlandson KM, Umbleja T, Lu MT, Taron J, Ribaudo HJ, Overton ET, Presti RM, Haas DW, Sax PE, Yin MT, Zhai BK, Louis R, Upadhyay N, Eslami P, Douglas PS, Zanni MV, Fitch KV, Fulda ES, Fichtenbaum CJ, Malvestutto CD, Grinspoon SK, Brown TT. Associations of Muscle Density and Area With Coronary Artery Plaque and Physical Function. J Acquir Immune Defic Syndr. 2023 Oct 1;94(2):174-184. doi: 10.1097/QAI.0000000000003244. PMID 37368931
- [Result] Abidi MZ, Umbleja T, Overton ET, Burdo T, Flynn JM, Lu MT, Taron J, Schnittman SR, Fitch KV, Zanni MV, Fichtenbaum CJ, Malvestutto C, Aberg JA, Fulda ES, Eckard AR, Manne-Goehler J, Tuan JJ, Ribaudo HJ, Douglas PS, Grinspoon SK, Brown TT, Erlandson KM. Cytomegalovirus IgG is Associated With Physical Function But Not Muscle Density in People With HIV. J Acquir Immune Defic Syndr. 2024 Apr 15;95(5):470-478. doi: 10.1097/QAI.0000000000003377. PMID 38180893
- [Result] Umbleja T, Brown TT, Overton ET, Ribaudo HJ, Schrack JA, Fitch KV, Douglas PS, Grinspoon SK, Henn S, Arduino RC, Rodriguez B, Benson CA, Erlandson KM. Physical Function Impairment and Frailty in Middle-Aged People Living With Human Immunodeficiency Virus in the REPRIEVE Trial Ancillary Study PREPARE. J Infect Dis. 2020 Jul 9;222(Suppl 1):S52-S62. doi: 10.1093/infdis/jiaa249. PMID 32645163
- [Derived] Erlandson KM, Umbleja T, Ribaudo HJ, Schrack JA, Overton ET, Fichtenbaum CJ, Fitch KV, Roa JC, Diggs MR, Wood K, Zanni MV, Bloomfield GS, Malvestutto C, Aberg JA, Rodriguez-Barradas MC, Morones RG, Breaux K, Douglas PS, Grinspoon SK, Brown TT. Pitavastatin Is Well-Tolerated With no Detrimental Effects on Physical Function. Clin Infect Dis. 2025 Feb 24;80(2):425-433. doi: 10.1093/cid/ciae422. PMID 39159048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from March 14, 2017 to February 6, 2019 at REPRIEVE U.S. sites participating in the REPRIEVE Mechanistic Substudy.
Period: Overall Study
Arm/Group | Pitavastatin | Placebo
Started | 316 | 286
Completed | 270 | 236
Not Completed | 46 | 50
Not completed — Lost to Follow-up | 34 | 27
Not completed — Withdrawal by Subject | 12 | 22
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin | Placebo | Total
Number analyzed (Participants) | 316 | 286 | 602
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [47 to 55] | 51 [47 to 55] | 51 [47 to 55]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity was reported by the participants.
  Participants
    Cisgender | 304 | 278 | 582
    Transgender spectrum | 5 | 6 | 11
    Not reported | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth.
  Participants
    Female | 65 | 46 | 111
    Male | 251 | 240 | 491
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the participants.
  Participants
    Hispanic or Latino | 56 | 52 | 108
    Not Hispanic or Latino | 257 | 232 | 489
    Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was reported by the participants. "Other" race includes participants who identified as native or indigenous to the enrollment region, as having more than one race, or as having an unknown race.
  Participants
    White | 160 | 153 | 313
    Black or African American | 126 | 112 | 238
    Asian | 3 | 2 | 5
    Other | 27 | 19 | 46
Region of Enrollment [Number; unit: participants]
  United States | 316 | 286 | 602
Enrollment cohort [Count of Participants; unit: Participants] — Enrollment cohort shows participants who enrolled into PREPARE concurrently with REPRIEVE (prospective enrollment) by co-enrollment in Mechanistic Substudy, and participants enrolled from REPRIEVE and Mechanistic Substudy within 24 months of their REPRIEVE enrollment (retrospective enrollment).
  Participants
    Prospective (Mechanistic Substudy) | 87 | 78 | 165
    Prospective (REPRIEVE only) | 60 | 43 | 103
    Retrospective (Mechanistic Substudy) | 169 | 165 | 334
CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — CD4 cell count at REPRIEVE enrollment (prior to initiating study treatment).
  cells/mm^3 | 615 [460 to 802] | 609 [445 to 785] | 609 [452 to 794]
HIV-1 RNA [Count of Participants; unit: Participants] — HIV-1 RNA at REPRIEVE enrollment (prior to initiating study treatment). HIV-1 RNA was captured if available through standard of care. Population: All participants enrolled with HIV-1 RNA result available through standard of care.
  Participants
    number analyzed (Participants) | 309 | 278 | 587
    <50 copies/mL | 288 | 262 | 550
    ≥50 copies/mL | 21 | 16 | 37
Chair rise rate [Mean (Standard Deviation); unit: rises per minute] — Chair rise rate at PREPARE entry calculated based on the time to complete 10 repeated chair stands. For participants enrolled into PREPARE retrospectively within 24 months of REPRIEVE enrollment, this may not represent physical function at the time of REPRIEVE entry. Population: All participants enrolled with chair stand test completed at PREPARE entry.
  rises per minute
    number analyzed (Participants) | 315 | 283 | 598
    (all) | 25.2 (7.6) | 25.0 (7.3) | 25.1 (7.5)
Gait speed [Mean (Standard Deviation); unit: meters per second] — Gait speed at PREPARE entry calculated based on the average of two 4-meter walk times. For participants enrolled into PREPARE retrospectively within 24 months of REPRIEVE enrollment, this may not represent physical function at the time of REPRIEVE entry. Population: All participants enrolled with 4-meter walk test completed at PREPARE entry.
  meters per second
    number analyzed (Participants) | 316 | 284 | 600
    (all) | 1.00 (0.21) | 1.00 (0.23) | 1.00 (0.22)
Grip strength [Mean (Standard Deviation); unit: kg] — Grip strength at PREPARE entry calculated as the average of three measurements on a handheld Jamar dynamometer. For participants enrolled into PREPARE retrospectively within 24 months of REPRIEVE enrollment, this may not represent physical function at the time of REPRIEVE entry. Population: All participants enrolled with grip strength test completed at PREPARE entry.
  kg
    number analyzed (Participants) | 311 | 283 | 594
    (all) | 34.3 (9.8) | 35.1 (9.9) | 34.7 (9.9)
Balance: Able to hold single-leg stand for 30 seconds [Count of Participants; unit: Participants] — Ability to hold single-leg-stand for 30 seconds at PREPARE entry. For participants enrolled into PREPARE retrospectively within 24 months of REPRIEVE enrollment, this may not represent physical function at the time of REPRIEVE entry. Population: All participants enrolled with balance test completed at PREPARE entry.
  Participants
    number analyzed (Participants) | 316 | 285 | 601
    Able to hold position | 246 | 222 | 468
    Not able to hold position | 70 | 63 | 133
Physical Function Impairment by SPPB score [Count of Participants; unit: Participants] — Impairment was classified as Short Physical Performance Battery (SPPB) score (≤10) and no impairment as score of 11-12 at PREPARE entry. For participants enrolled into PREPARE retrospectively within 24 months of REPRIEVE enrollment, this may not represent physical function at the time of REPRIEVE entry. Population: All participants enrolled with physical performance tests (repeated chair stands, 4-meter walk, balance) completed at PREPARE entry.
  Participants
    number analyzed (Participants) | 316 | 284 | 600
    Impairment | 104 | 111 | 215
    No impairment | 212 | 173 | 385
Modified SPPB score [Mean (Standard Deviation); unit: units on a scale] — mSPPB score (ranging from 0-unable to perform to 3-maximal performance) at PREPARE entry calculated as a sum of the following components each divided by the maximal possible performance: (1) chair rise rate (stands/second) divided by maximal performance of one stand/second; (2) proportion of total standing balance time calculated as the total time each of the semi-tandem, tandem and one-leg stand positions were held (maximum 30 seconds each) divided by 90 seconds; and (3) gait speed (meters/second) based on average of the 4-meter walk results divided by maximal performance of 2 meters/second. Population: All participants enrolled with physical function tests (repeated chair stands, 4-meter walk, balance) completed at PREPARE entry.
  units on a scale
    number analyzed (Participants) | 316 | 284 | 600
    (all) | 1.86 (0.24) | 1.86 (0.27) | 1.86 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Physical Function: Rate of Change in Chair Rise Rate
Description: Chair rise rate was calculated as the number of chair stands performed divided by the time to complete 10 chair stands. Participants unable to attempt the test were assigned the worst time (9 seconds/stand for every stand not done). Linear mixed effects models for repeated measures were used to estimate annualized rate of change (slope), and the difference between treatment groups (interaction between slope and treatment group). Negative annualized rate of change reflects decline over time, positive improvement over time.
Time Frame: Entry and months 12, 24, 36, 48, 60
Population: All participants enrolled with any chair rise rate data available.
Measure: Mean (95% Confidence Interval); unit: rises/minute per year
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
rises/minute per year | -0.035 [-0.20 to 0.13] | 0.07 [-0.11 to 0.24]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.31, Mixed Models Analysis; P-value is from the time and treatment group interaction; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.30 to 0.10] — Treatment effect was estimated as the difference in annualized rate of change (slope) with randomized pitavastatin compared to placebo from linear mixed effects models (0 reflects no difference between treatment groups)

2. Primary Outcome: Mechanistic: Rate of Change in Inflammatory Index Score (IIS)
Description: Conditional on the positive findings on the primary physical function, the IIS score will be calculated as 1/3 log [interleukin-6 (IL-6)] + 2/3 log [soluble tumor necrosis factor receptor 1 (sTNFR-1)] using specimens collected as part of the main study REPRIEVE, and used to evaluate mechanistic pathways through which pitavastatin affects physical function.
Time Frame: Baseline and 12 months
Population: The specimen testing was not performed.
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Muscle Quality: Paraspinal Muscle Density
Description: Paraspinal muscle (a back muscle) density was measured in Hounsfield units (HU, lower values indicate fattier muscle) from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE. HU are used to measure the radiation attenuation of muscle in CT scans. Muscle tissue was identified as voxels with attenuation of -190 HU (very low density muscle, the fattiest) to 100 HU (high density muscle, the leanest).
Time Frame: Baseline and 24 months
Population: Participants who remained on study treatment at Month 24 (per-protocol set) and had data for this outcome available at both baseline and month 24.
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 254 | 255
HU
  Baseline | 36.8 (18.1) | 36.4 (16.7)
  Month 24 | 36.2 (16.7) | 35.4 (18.1)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.62, Regression, Linear; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-1.72 to 2.88] — Treatment group difference was estimated using baseline-adjusted linear regression model

4. Secondary Outcome: Physical Function: Rate of Change in Gait Speed
Description: Gait speed was calculated as 4 meters divided by the average time to complete the 4-meter walk. Participants unable to attempt the test were assigned the worst gait speed (0 meters/second). Linear mixed effects models for repeated measures were used to estimate annualized rate of change (slope), and the difference between treatment groups (interaction between slope and treatment group). Negative annualized rate of change reflects decline over time, positive improvement over time.
Time Frame: Entry and months 12, 24, 36, 48 and 60.
Population: All participants enrolled with any gait speed data available.
Measure: Mean (95% Confidence Interval); unit: meters/second per year
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
meters/second per year | -0.013 [-0.018 to -0.008] | -0.012 [-0.017 to -0.007]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.61, Mixed Models Analysis; P-value is from the time and treatment group interaction; Mean Difference (Net) = -0.001, 95% CI 2-sided [-0.007 to 0.004] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Physical Function: Rate of Change in Grip Strength
Description: Grip strength was calculated as the average of three measurements in the dominant hand by Jamar Hydraulic Hand Dynamometer. Participants unable to attempt the test were assigned the worst result (0 kg). Linear mixed effects models for repeated measures were used to estimate annualized rate of change (slope), and the difference between treatment groups (interaction between slope and treatment group). Negative annualized rate of change reflects decline over time, positive improvement over time.
Time Frame: Entry and months 12, 24, 36, 48 and 60
Population: All participants enrolled with any grip strength data available.
Measure: Mean (95% Confidence Interval); unit: kg per year
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
kg per year | -0.39 [-0.57 to -0.21] | -0.36 [-0.56 to -0.17]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.80, Mixed Models Analysis; P-value is from the time and treatment group interaction; Mean Difference (Net) = -0.028, 95% CI 2-sided [-0.25 to 0.19] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Physical Function: Rate of Change in Risk of Impairment According to Balance
Description: Physical function impairment according to balance was defined as inability to hold single-leg stand for 30 seconds. Annualized risk of impairment year-over-year (ratio of risk per year, compared to risk per previous year) was estimated using log-binomial regression models for repeated data using GEE (relative risk of >1 reflects an increase in risk compared to previous year, relative risk <1 a decrease in risk compared to previous year). GEE (generalized estimating equations) is a statistical method for analyzing repeated measures, such as measurements of the outcome in participants at multiple time points.
Time Frame: Entry and months 12, 24, 36, 48, 60
Population: All participants enrolled with any balance data available.
Measure: Mean (95% Confidence Interval); unit: ratio per year
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
ratio per year | 1.08 [1.04 to 1.12] | 1.06 [1.02 to 1.10]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.33, Log-binomial regression using GEE; P-value is from the time and treatment group interaction; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.98 to 1.06] — Treatment effect is shown as relative annualized risk of impairment in the pitavastatin group compared to placebo (1 reflects no difference between treatment groups)

7. Secondary Outcome: Physical Function: Rate of Change in Modified SPPB Score
Description: Modified SPPB score (on scale from 0-worst to 3-best) was calculated as a sum of the following components each divided by the maximal possible performance: (1) chair rise rate (stands/second) divided by maximal performance of one stand/second; (2) proportion of total standing balance time calculated as the total time each of the semi-tandem, tandem and one-leg stand positions were held (maximum 30 seconds each) divided by 90 seconds; and (3) gait speed (meters/second) based on average of the 4-meter walk results divided by maximal performance of 2 meters/second. Linear mixed effects models for repeated measures were used to estimate annualized rate of change (slope), and the difference between treatment groups (interaction between slope and treatment group). Negative annualized rate of change reflects decline over time, positive improvement over time.
Time Frame: Entry and months 12, 24, 36, 48 and 60
Population: All participants enrolled with any mSPPB data available.
Measure: Mean (95% Confidence Interval); unit: score on a scale per year
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
score on a scale per year | -0.019 [-0.026 to -0.013] | -0.014 [-0.021 to -0.007]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.18, Mixed Models Analysis; P-value is from the time and treatment group interaction; Mean Difference (Net) = -0.005, 95% CI 2-sided [-0.013 to 0.002] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Physical Function: Rate of Change in Risk of Impairment According to SPPB
Description: Physical function impairment according to composite Short Physical Performance Battery (SPPB, consisting of repeated chair stands, balance and gait speed tests) was defined as score <=10. In the absence of trend over time, average relative risk of impairment over follow-up time (ratio) was estimated using log-binomial regression models for repeated data using GEE (relative average risk of >1 reflects an increase in risk over follow-up time, relative average risk <1 a decrease in risk over follow-up time). GEE (generalized estimating equations) is a statistical method for analyzing repeated measures, such as measurements of the outcome in participants at multiple time points.
Time Frame: Entry and months 12, 24, 36, 48, 60
Population: All participants enrolled with any SPPB data available.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
ratio | 1.00 [0.82 to 1.22] | 0.95 [0.77 to 1.16]
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Test type: Superiority; p = 0.47, Log-binomial regression using GEE; P-value is from the time (before vs. after study treatment initiation) and treatment group interaction; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.91 to 1.24] — Treatment effect is shown as relative average risk of impairment over follow-up time in the pitavastatin group compared to placebo (1 reflects no difference between treatment groups)

9. Secondary Outcome: Physical Function: Impairment According to DASI
Description: Impairment was classified according to self-administered Duke Activity Status Index questionnaire score (on scale from 0-worst to 58.2-best) as no impairment (the max score of 58.2), some impairment (score of 34.7-<58.2), moderate impairment (9.95-<34.7) and severe impairment (0-<9.95).
Time Frame: Baseline, month 24 and end of REPRIEVE (average at 5.6 years)
Population: All participants enrolled with DASI questionnaire completed at the given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
Participants
  Baseline: No impairment | 219 | 192
  Baseline: Some impairment | 74 | 66
  Baseline: Moderate impairment | 23 | 26
  Baseline: Severe impairment | 0 | 1
  Month 24: number analyzed (Participants) | 280 | 254
  Month 24: No impairment | 165 | 159
  Month 24: Some impairment | 84 | 71
  Month 24: Moderate impairment | 31 | 22
  Month 24: Severe impairment | 0 | 2
  End of REPRIEVE: number analyzed (Participants) | 249 | 226
  End of REPRIEVE: No impairment | 135 | 129
  End of REPRIEVE: Some impairment | 77 | 64
  End of REPRIEVE: Moderate impairment | 37 | 28
  End of REPRIEVE: Severe impairment | 0 | 5

10. Secondary Outcome: Frailty Phenotype
Description: Frailty Phenotype was defined based on the following components: (1) weight loss (self-report of unintentional weight loss of 10 or more pounds in the prior year), (2) exhaustion (experiencing at least three to four times per week the feeling that "everything I do is an effort" or "sometimes I cannot get going", (3) low physical activity (being "limited a lot" in response to the Short Form 36 question "does your health limit you in vigorous activities such as running, lifting heavy objects, or participating in strenuous sports?", (4) slow gait by average of two 4-meter walk times, and (5) weak grip by average of three measurements on a handheld Jamar dynamometer. Participants were classified as non-frail if they had no components present, pre-frail with one or two components present, and frail with three or more components present.
Time Frame: Entry and months 12, 24, 36, 48, 60
Population: All participants enrolled with frailty phenotype data available. (Data availability at baseline and 12 depends on timing of PREPARE enrollment relative to REPRIEVE enrollment.)
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
Participants
  Baseline: number analyzed (Participants) | 144 | 120
  Baseline: Non-frail | 74 | 65
  Baseline: Pre-frail | 65 | 45
  Baseline: Frail | 5 | 10
  Month 12: number analyzed (Participants) | 181 | 156
  Month 12: Non-frail | 89 | 72
  Month 12: Pre-frail | 82 | 74
  Month 12: Frail | 10 | 10
  Month 24: number analyzed (Participants) | 252 | 218
  Month 24: Non-frail | 113 | 99
  Month 24: Pre-frail | 124 | 105
  Month 24: Frail | 15 | 14
  Month 36: number analyzed (Participants) | 226 | 200
  Month 36: Non-frail | 102 | 104
  Month 36: Pre-frail | 114 | 86
  Month 36: Frail | 10 | 10
  Month 48: number analyzed (Participants) | 239 | 204
  Month 48: Non-frail | 108 | 109
  Month 48: Pre-frail | 112 | 84
  Month 48: Frail | 19 | 11
  Month 60: number analyzed (Participants) | 231 | 204
  Month 60: Non-frail | 95 | 93
  Month 60: Pre-frail | 114 | 101
  Month 60: Frail | 22 | 10

11. Secondary Outcome: Physical Activity: Frequency of <30 Minutes of Physical Activity 3 or More Days a Week
Description: Self-reported physical activity evaluated by the questionnaire "Rapid Eating and Activity Assessment for Patients" (REAP) question 27: In an average week, how often do you do <30 minutes of physical activity 3 or more days a week?
Time Frame: Baseline and months 12, 24, 36, 48, 60
Population: All participants enrolled with REAP Question 27 data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
Participants
  Baseline: number analyzed (Participants) | 315 | 285
  Baseline: Rarely/never | 140 | 137
  Baseline: Sometimes | 92 | 82
  Baseline: Usually/often | 83 | 66
  Month 12: number analyzed (Participants) | 200 | 177
  Month 12: Rarely/never | 119 | 89
  Month 12: Sometimes | 30 | 43
  Month 12: Usually/often | 51 | 45
  Month 24: number analyzed (Participants) | 278 | 246
  Month 24: Rarely/never | 124 | 108
  Month 24: Sometimes | 76 | 80
  Month 24: Usually/often | 78 | 58
  Month 36: number analyzed (Participants) | 219 | 201
  Month 36: Rarely/never | 108 | 113
  Month 36: Sometimes | 52 | 37
  Month 36: Usually/often | 59 | 51
  Month 48: number analyzed (Participants) | 232 | 202
  Month 48: Rarely/never | 111 | 110
  Month 48: Sometimes | 51 | 38
  Month 48: Usually/often | 70 | 54
  Month 60: number analyzed (Participants) | 221 | 185
  Month 60: Rarely/never | 115 | 100
  Month 60: Sometimes | 42 | 36
  Month 60: Usually/often | 64 | 49

12. Secondary Outcome: Physical Activity: Frequency of Watching >2 Hours of TV or Videos a Day
Description: Self-reported physical activity evaluated by the questionnaire "Rapid Eating and Activity Assessment for Patients" (REAP) question 28: In an average week, how often do you do watch >2 hours of TV or videos a day?
Time Frame: Baseline and months 12, 24, 36, 48, 60
Population: All participants enrolled with REAP Question 28 data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 316 | 285
Participants
  Baseline: number analyzed (Participants) | 313 | 284
  Baseline: Rarely/never | 67 | 48
  Baseline: Sometimes | 88 | 92
  Baseline: Usually/often | 158 | 144
  Month 12: number analyzed (Participants) | 200 | 177
  Month 12: Rarely/never | 53 | 42
  Month 12: Sometimes | 55 | 46
  Month 12: Usually/often | 92 | 89
  Month 24: number analyzed (Participants) | 277 | 246
  Month 24: Rarely/never | 58 | 59
  Month 24: Sometimes | 84 | 87
  Month 24: Usually/often | 135 | 100
  Month 36: number analyzed (Participants) | 219 | 201
  Month 36: Rarely/never | 52 | 46
  Month 36: Sometimes | 58 | 54
  Month 36: Usually/often | 109 | 101
  Month 48: number analyzed (Participants) | 232 | 202
  Month 48: Rarely/never | 54 | 45
  Month 48: Sometimes | 54 | 56
  Month 48: Usually/often | 124 | 101
  Month 60: number analyzed (Participants) | 221 | 185
  Month 60: Rarely/never | 55 | 32
  Month 60: Sometimes | 45 | 41
  Month 60: Usually/often | 121 | 112

13. Secondary Outcome: Muscle Quality: Pectoral Muscle Density
Description: Pectoral (a chest muscle) density was measured in Hounsfield units (HU) from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE.
Time Frame: Baseline and month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 253 | 252
HU
  Baseline | 41.4 (15.9) | 40.9 (16.2)
  Month 24 | 41.5 (16.1) | 41.8 (15.4)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.55, Regression, Linear; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.7 to 1.4] — Treatment group difference at Month 24 (pitavastatin minus placebo) was estimated using baseline-adjusted linear regression model (0 reflects no difference between treatment groups)

14. Secondary Outcome: Muscle Quality: Infraspinatus Muscle Density
Description: Infraspinatus (an upper back muscle) density was measured in Hounsfield units (HU) from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE.
Time Frame: Baseline and month 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: HU
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 237 | 234
HU
  Baseline | 44.3 (17.1) | 42.6 (18.1)
  Month 24 | 44.2 (13.4) | 44.0 (15.6)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.67, Regression, Linear; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.8 to 1.8] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Muscle Area: Paraspinal Muscle Area
Description: Paraspinal muscle (a back muscle) area was measured from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE.
Time Frame: Baseline and month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2/m
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 254 | 255
cm^2/m
  Baseline | 12.0 (4.8) | 12.5 (5.1)
  Month 24 | 12.1 (4.6) | 12.5 (4.9)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.98, Regression, Linear; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.50 to 0.52] — Treatment group difference (pitavastatin minus placebo) at Month 24 was estimated using baseline-adjusted linear regression model (0 reflects no difference between treatment groups)

16. Secondary Outcome: Muscle Area: Pectoral Muscle Area
Description: Pectoral muscle (a chest muscle) area was measured from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE.
Time Frame: Baseline and month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2/m
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 253 | 252
cm^2/m
  Baseline | 8.3 (5.4) | 8.6 (5.1)
  Month 24 | 8.2 (4.9) | 8.7 (5.2)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.31, Regression, Linear; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.3] — [estimate comment as in outcome 13, analysis 1]

17. Secondary Outcome: Muscle Area: Infraspinatus Muscle Area
Description: Infraspinatus muscle (an upper back muscle) area was measured from central reading of CT scans performed as part of A5333s, the Mechanistic Substudy of REPRIEVE.
Time Frame: Baseline and month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2/m
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 237 | 234
cm^2/m
  Baseline | 6.3 (4.5) | 6.3 (4.6)
  Month 24 | 6.5 (4.6) | 6.2 (4.2)
Statistical Analysis 1: Comparison: Pitavastatin vs Placebo; Comparison of Month 24 values; Test type: Superiority; p = 0.21, Regression, Linear; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 0.9] — [estimate comment as in outcome 13, analysis 1]

18. Secondary Outcome: Mechanistic: Serum Concentrations of Biomarkers
Description: Conditional on the positive findings on the primary physical function, select biomarkers including each individual biomarker of the IIS (IL-6, sTNFR-1) as well as other biomarkers implicated in the pathogenesis of physical function impairment or those that may mediate the effects of statins on systemic inflammation will be used to evaluate mechanistic pathways through which pitavastatin affects physical function. The specific list of biomarkers of interest will be finalized closer to the time of analysis, incorporating the developments in the field over the few years from study development to completion.
Time Frame: Baseline and month 12
Population: The specimen testing was not done.
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: For all-cause mortality: from entry to Month 60
Description: There was no adverse event data collection in PREPARE.
Arm/Group | Pitavastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 7/316 | 10/286
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03070223/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03070223/SAP_001.pdf